CLINICAL TRIAL: NCT02487407
Title: Effects of ODM-109 on Respiratory Function in Patients With ALS. A Randomized, Double Blind, Placebo-controlled, Cross-over, 3-period, Multicenter Study With Open-label Follow-up Extension
Brief Title: Effects of ODM-109 on Respiratory Function in Patients With Amyotrophic Lateral Sclerosis
Acronym: ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3119001
Record Dates: First submitted 2015-06-08; First posted 2015-07-01 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2016-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ODM-109 (Experimental): ODM-109 capsules for oral administration
  Interventions: Drug: ODM-109; Drug: Placebo for ODM-109
- Placebo for ODM-109 (Placebo Comparator): Placebo ODM-109 capsules for oral administration
  Interventions: Drug: ODM-109; Drug: Placebo for ODM-109

INTERVENTIONS:
Drug: ODM-109 — ODM-109 1 mg capsule for oral administration.
  Other Names: Levosimendan
Drug: Placebo for ODM-109 — Placebo capsule for oral administration.
  Other Names: Placebo for Levosimendan

SUMMARY:
In the double-blind, cross-over part of the study, ODM-109 capsules and placebo capsules for ODM-109 will be administered for 2 weeks separated by a 19-23 days wash-out period. During each treatment period of the double-blind cross-over part, there will be a baseline visit (day 1) and 2 visits (5 ± 2 and 14 ± 2 days) after the start of study treatment. After completing the 3rd treatment period, the subjects will continue in the open-label follow-up part for 6 months. During the open-label follow-up, visits will be at 1, 3 and 6 months. An end-of-study visit will take place 14-25 days after the last study treatment administration for each subject. The study duration will be about 13-14 weeks for the double-blind cross-over part, and about 9-10 months for the entire study including the 6 months open-label follow-up.

The number of randomised study subjects is planned to be approximately 54 in cross-over comparison. The maximum number of subjects will not exceed 70.

Primary objective is to investigate the efficacy of oral ODM-109 on respiratory function in patients with amyotrophic lateral sclerosis (ALS).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) for participation in the study will be obtained from the subject (or from the subject's next of kin, caregiver, or other legally acceptable representative in case the study subject him/herself cannot sign the IC due to severe muscle weakness).
* Age of at least 18 years.
* Male or female subjects with diagnosis of laboratory supported probable, probable or definite ALS according to El Escorial revised criteria (Brooks BR et al., 2000). Full electromyogram (EMG) report available compatible with ALS according to an experienced neurophysiologist.
* Ability to swallow the study treatment capsules.
* An upright (sitting position) SVC between 60-90% of the predicted value for age, height and sex at screening visit.
* Normal oxygen saturation during daytime (measure of ≥ 95% when steady state has been reached with a reliable read) in sitting position measured by pulse oximetry.
* Disease duration from symptom onset (defined by first muscle weakness or dysarthria) of 12-48 months.
* Using riluzole. The dose must have been stable for at least 4 weeks prior to screening at a dose of 50 mg b.i.d.

Exclusion Criteria:

* Subject in whom other causes of neuromuscular weakness have not been excluded.
* Subject with a diagnosis of another neurodegenerative disease (e.g. Parkinson's or Alzheimer's disease).
* Assisted ventilation or gastrostomy of any type during the preceding 3 months prior to screening or predicted to be required within the randomised, double-blind cross-over part of the study.
* Recorded diagnosis or evidence of major psychiatric diagnosis, significant cognitive impairment or clinically evident dementia.
* Any major surgery within 1 month before the screening visit or patients who are scheduled for any major surgery during the planned study period.
* Potassium < 3.7 mmol/l or > 5.5 mmol/l at screening.
* Creatinine > 170 μmol/l at screening or on dialysis.
* Blood haemoglobin < 10 g/dl at screening.
* Clinically significant hepatic impairment at the discretion of the investigator.
* Women of reproductive age without a negative pregnancy test and without a commitment to using an acceptable method of barrier or hormonal contraception (e.g. condoms, diaphragms, oral contraceptives and long acting progestin agents), if sexually active during the study, and for 1 month after the last dose of the study treatment. Women who are postmenopausal (1 year since last menstrual cycle), surgically sterilised or who have undergone a hysterectomy are considered not to be reproductive and can be included.
* Known hypersensitivity to levosimendan.
* Administration of levosimendan within 30 days prior to screening visit.
* Patients with history of botulinum toxin treatment for any reason.
* Patients with known history of human immunodeficiency virus infection.
* History of significant arrhythmias or other cardiac events
* Any other clinically significant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, neurological or psychiatric disorder or any other major concurrent illness that in the opinion of the investigator could interfere with the interpretation of the study results or constitute a health risk for the subject if he/she took part in the study.
* Blood donation or loss of significant amount of blood within 60 days prior to screening.
* Participation in a clinical trial with any experimental treatment within 30 days prior to the screening visit or previous participation in the present study.
* Any other condition that in the opinion of the investigator could interfere with the interpretation of the study results or constitute a health risk for the subject if he/she took part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Slow vital capacity SVC | 9 months
  Pulmonary assessment

SECONDARY OUTCOMES:
Hand grip strength and submaximal hand grip strength endurance | 3 months
  Assessment
Changes in subject's clinical condition (relative to the baseline/day 1 of the given treatment period) will be assessed using the Clinical Global Impression of Change (CGI-C) | 3 months
  Scales
Quality of life | 9 months
  Questionnaire
Revised ALS Functional Rating Scale ALSFRS-R | 9 months
  Scale
Oxygen saturation | 9 months
  Assessment
The concentrations of ODM-109, OR-1855 and OR-1896 | 3 months
  Pharmacokinetics Blood samples.
Determination of subject's acetylation status | 1 day (once at baseline)
  Pharmacogenomics Blood samples.
Sniff nasal pressure SNP | 9 months
  SNP will be assessed in sitting position. SNP will be performed for 10 times. The highest value (cmH2O) measured will be the SNP variable.
Fatigue assessment | 3 months
  Visual analogue Scale VAS

CONTACTS AND LOCATIONS:
Overall Officials: Merja Mäkitalo, CSD, Study Director — Finland
Locations (11):
- Germany (4):
  - Charite Universitatsmedizin Berlin, Berlin
  - Medical School Hannover, Hanover
  - University Clinical Jena, Jena
  - University Hospital of Ulm, Ulm
- Beaumont Hospital, Dublin, Ireland
- University Medical Centre Utrecht, Utrecht, Netherlands
- United Kingdom (5):
  - Royal Sussex County Hospital, Brighton
  - The Walton Centre, Liverpool
  - London Kings College Hospital, London
  - Royal London Hospital, London
  - University of Sheffield, Sheffield

REFERENCES:
- [Derived] Al-Chalabi A, Shaw P, Leigh PN, van den Berg L, Hardiman O, Ludolph A, Aho VV, Sarapohja T, Kuoppamaki M. Oral levosimendan in amyotrophic lateral sclerosis: a phase II multicentre, randomised, double-blind, placebo-controlled trial. J Neurol Neurosurg Psychiatry. 2019 Oct;90(10):1165-1170. doi: 10.1136/jnnp-2018-320288. Epub 2019 Jul 17. PMID 31315908